CLINICAL TRIAL: NCT05103553
Title: Value Based Health Care in Systemic Sclerosis: What is the Optimal Follow-up for Patients With Systemic Sclerosis?
Brief Title: What is the Optimal Follow-up for Patients With Systemic Sclerosis?
Acronym: PRASSc
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Jeska K. de Vries-Bouwstra, Dr. / Principal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P21.069
Record Dates: First submitted 2021-10-11; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Systemic Sclerosis
Keywords: Prediction model; Systemic Sclerosis; Value based health care
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Ambulatory Care Facilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Annual screening at outpatient clinic (Experimental): After signing informed consent, patients with low risk for disease progression (in the low or intermediate risk group) wil be randomized into the intervention group (annual assessment at the outpatient clinic). Due to the nature of the intervention, the randomization will not be blinded, as this is not possible.
  Interventions: Other: Outpatient Clinic
- Annual screening at Care Pathway Systemic Sclerosis (No Intervention): After signing informed consent, patients with low risk for disease progression (in the low or intermediate risk group) will be randomized into the control group (annual assessment at the care pathway). Due to the nature of the intervention, the randomization will not be blinded, as this is not possible.

INTERVENTIONS:
Other: Outpatient Clinic — Follow-up in outpatient clinic
  Arms: Annual screening at outpatient clinic

SUMMARY:
Systemic sclerosis (SSc) is a complex multisystem rheumatic autoimmune disease. Currently, evidence based guidelines for frequency and intensity of follow-up of SSc patients are not available. Based on expert consensus annual extensive evaluation is recommended. To provide comprehensive multidisciplinary care integrated with evaluation of organ involvement and as such, reducing health care utilization while improving the quality of care for the patient, the "Leiden Combined Care in SSc (CCISS) pathway" was started in 2009. Data collected on disease progression in the patients that participate in this care pathway show that 50% of the patients have relatively mild disease, without any disease progression over time. Therefore there is a need for tailor made care in SSc patients in accordance to disease activity. To enable this, a prediction model was developed that can identify patients with low risk for disease progression.

DETAILED DESCRIPTION:
Objectives: To evaluate in SSc patients with low risk for disease progression 1) whether assessment in an outpatient clinic setting is an acceptable alternative for evaluation in the Care Pathway. Outcome parameters we will evaluate include 1) health care utilization, 2) patients' perception of the disease and delivery of care, 3) health-related quality of life and 4) disease progression. Health care utilization as primary outcome is defined as number of contacts with heath care providers during 12 months.

Study population: Patients with a clinical diagnosis of SSc that participated in the Combined Care in Systemic Sclerosis cohort from Leiden University Medical Center (LUMC), or in the comparable care pathway of the Haga hospital and Haaglanden Medical Center (HMC), and that have had at least two care pathway evaluations are eligible to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Participation in the prospective Haga, HMC or LUMC cohort
2. Clinical diagnosis of SSc
3. Age of ≥18 years
4. >= two evaluations in the Care Pathway
5. Low or intermediate risk for disease progression according to the prediction model
6. Written informed consent

Exclusion Criteria:

1. Patients with SSc who are part of ongoing (randomized) trials
2. Patients who have had an autologous stem cell transplantation in the past five years
3. Patients with SSc who were categorized as high risk for disease progression according to the prediction model.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Health care utilization Baseline | Baseline
  Includes different health-care services: rheumatologist, other medical specialists, General Practioner (GP), health professionals, hospital admission, hospital based day-care. Number of contacts/visits within previous 6 months will be counted.
Health care utilization after 6 months | 6 months
  Includes different health-care services: rheumatologist, other medical specialists, General Practioner (GP), health professionals, hospital admission, hospital based day-care. Number of contacts/visits within previous 6 months will be counted.
Health care utilization after 12 months | 12 months
  Includes different health-care services: rheumatologist, other medical specialists, General Practioner (GP), health professionals, hospital admission, hospital based day-care. Number of contacts/visits within previous 6 months will be counted.
Health care utilization after 18 months | 18 months
  Includes different health-care services: rheumatologist, other medical specialists, General Practioner (GP), health professionals, hospital admission, hospital based day-care. Number of contacts/visits within previous 6 months will be counted.
Health care utilization after 24 months | 24 months
  Includes different health-care services: rheumatologist, other medical specialists, General Practioner (GP), health professionals, hospital admission, hospital based day-care. Number of contacts/visits within previous 6 months will be counted.

SECONDARY OUTCOMES:
Disease progression | Baseline, 6 months, 12 months, 18 months, 24 months
  Defined as progression in different organ systems.
health-related quality of life using 36-item short form survey (SF-36) | Baseline, 6 months, 12 months, 18 months, 24 months
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. Rely upon patient self-reporting.
health-related quality of life using EuroQol 5D (EQ5D) | Baseline, 6 months, 12 months, 18 months, 24 months
  comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. each dimension has 5 levels varying from no problems until extreme problems. Each answer results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.The EQ visual analogue scale (VAS) records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's judgement.
Illness perception using the validated instrument Brief Illness Perception Questionnaire (BIPQ ) | Baseline, 6 months, 12 months, 18 months, 24 months
  A nine-item scale designed to rapidly assess the cognitive and emotional representations of illness. Each question is be answered with a number on a scale of 0 until 10.

CONTACTS AND LOCATIONS:
Overall Officials: Jeska de Vries-Bouwstra, MD PhD, Principal Investigator — Leiden University Medical Center

IPD SHARING:
Plan to Share IPD: No